CLINICAL TRIAL: NCT05731830
Title: Takotsubo Syndrome and Air Pollution: the "Tako-Air" Study
Brief Title: Takotsubo Syndrome and Air Pollution
Acronym: Tako-Air
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MONTONE ROCCO ANTONIO, IRCCS Researcher, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5290
Record Dates: First submitted 2023-01-27; First posted 2023-02-16 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Takotsubo Syndrome
Keywords: Air Pollution; Takotsubo Syndrome; Stress cardiomyopathy
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Takotsubo Syndrome: Patients admitted to the Department of Cardiovascular Sciences of Fondazione Policlinico Universitario A. Gemelli IRCCS with a diagnosis of TTS. TTS will be diagnosed based on the most recent InterTAK Diagnostic Criteria. Myocarditis will be excluded based on clinical presentation (e.g.: previous flu-like symptoms, increased inflammatory biomarkers) and confirmed by cardiac magnetic resonance. We will further include all patients with a confirmed TTS diagnosis made between January 2016 and end of October 2022 (hypothetical beginning of prospective phase).
  Interventions: Other: Data extraction; Other: Clinical follow-up

INTERVENTIONS:
Other: Data extraction — The exposure of patients to air pollution compounds in the two years prior to the occurrence of TTS will be analysed. We will investigate: PM10, PM2.5, O3, NO2, C6H6, SO2 e CO. Residential addresses will be obtained from medical records. Annual average 24-h of pollutants levels will be measured matching each individual's home address, and the "ArpaLazio" website (http://www.arpalazio.net/main/aria/sci/basedati/chimici/chimici.php), which provides the concentration of NO, NO2, NOx, PM10, PM2.5, O3, CO, C6H6, SO2 expressed in micrograms per cubic meter (µg/m3). Hourly data are available for all gaseous pollutants, while the levels of PM10 and PM2.5 are expressed daily. Data will be obtained from the air quality monitor closest to each participant's residence that was active for the entire year, and short-term (daily and weekly) and long-term (annual) air pollution exposure will be quantified as daily, weekly, and annual average 24-h pollutants level of measurements before TTS.
Other: Clinical follow-up — All patients will undergo a clinical follow-up by telephonic interview and/or clinical visit at 6, 12, 24, 36, 48 and 60 months from hospital discharge, during which the incidence of MACE, defined as the composite of all-cause mortality, non-fatal MI, transient ischemic attack (TIA)/stroke, and hospitalization for heart failure, and the recurrence of TTA in the past months will be investigated and collected.

SUMMARY:
Takotsubo syndrome (TTS) is an acute and reversible form of myocardial injury characterized by typical regional wall motion abnormalities in the absence of culprit epicardial coronary artery disease frequently precipitated by significant emotional stress or serious physical illness. The clinical presentation is usually similar to acute myocardial infarction (MI), with chest pain and/or dyspnea, ST-segment elevation or depression and/or T-wave inversion on the resting electrocardiogram (ECG) and elevation of serum cardiac troponin. Although previously considered a benign disease, it is now clear that TTS is associated with severe acute complications during the acute phase including hemodynamic and electrical instability and up to 5% of in-hospital mortality.

The pathogenetic mechanisms of air pollution are likely to predispose to the occurrence as well as to mediate a worse clinical presentation and outcome of TTS, proving air pollution as a TTS risk factor.

DETAILED DESCRIPTION:
Background

Takotsubo syndrome (TTS) is an acute and reversible form of myocardial injury characterized by typical regional wall motion abnormalities in the absence of culprit epicardial coronary artery disease frequently precipitated by significant emotional stress or serious physical illness. The clinical presentation is usually similar to acute myocardial infarction (MI), with chest pain and/or dyspnea, ST-segment elevation or depression and/or T-wave inversion on the resting electrocardiogram (ECG) and elevation of serum cardiac troponin. Although previously considered a benign disease, it is now clear that TTS is associated with severe acute complications during the acute phase including hemodynamic and electrical instability and up to 5% of in-hospital mortality.

Notably, despite substantial research, the risk factors and pathophysiological mechanisms of TTS are not completely understood, with several hypotheses proposed but none offering a comprehensive explanation. Catecholamine-induced myocardial injury is likely to play a central role, as an emotionally or physically triggering event precipitating the syndrome can be identified in most cases and TTS has been associated with conditions of catecholamine excess (e.g.: pheochromocytoma, central nervous system disorders) and activated specific cerebral regions. Similarly, a markedly reduced parasympathetic activity has been reported during the acute phase of TTS. Moreover, recent studies reported abnormalities in both the functional structure and activity in the areas of the brain related to both emotions and the sympathetic nervous system including the basal ganglia, the hippocampus, the amygdala, and the insula, supporting the role of limbic system dysfunction as a potential mechanism in patients with TTS. Furthermore, it has been proposed that the impaired cardiac function could be the result of an acute coronary microvascular dysfunction with impaired microvascular perfusion leading to a demand-supply mismatch and an ischemic stunning. Therefore, the risk factors for endothelial dysfunction would predispose to the occurrence of TTS.

Air pollution is a complex mixture of unwanted particulate and gaseous material released into the environment by human activities and the world's fourth leading cause of disease and death. Of interest, accumulating evidence supports a consistent relationship between increased exposure to air pollution and CV diseases such as MI and heart failure. Urban ambient air pollution, in particular combustion-derived PM, has received the greatest scientific attention due to the high density of urban populations and increasing levels of traffic-derived emissions and urbanization of societies worldwide. PM includes both organic and inorganic particles (e.g.: dust, pollen, soot, smoke, liquid droplets) and is categorized according to the aerodynamic diameter into coarse particles (2.5-10 μm in diameter; PM10), fine particles (<2.5 μm in diameter; PM2.5), and ultrafine particles (<0.1 μm in diameter; PM0.1). The smallest particles, such as PM2.5 and PM0.1, may contribute disproportionately to the CV toxic effects due to their large reactive surface area and their ability to penetrate deeply into the alveoli and potentially directly into the bloodstream, causing damage and dysfunction of various tissues and cells far from the lung. Gaseous pollutants, in particular nitric dioxide (NO2), ozone (O3), carbon monoxide (CO) and sulphur dioxide (SO2), have been linked to increased morbidity and mortality from CV diseases, likely in an additive manner to PM2.5, but data are still scarce and frequently inconsistent. Mechanistically, the pathogenetic mechanism of air pollution toxicity on the CV system includes oxidative stress, systemic and vascular inflammation, endothelial dysfunction, autonomic and neuroendocrine disruption, metabolic alterations, transcriptional and epigenetic reprogramming. Furthermore, the acute responses to short-term (hours) air pollution exposure include sympathoadrenal activation, release of circulating inflammatory biomarkers, alterations of endothelial function, and acute vascular modifications, such as arterial vasoconstriction and impaired vascular reactivity. The acute effects of air pollution are even more significant in the context of chronic long-term (years) exposure. Indeed, chronic air pollution exposure, by promoting the development of a vulnerable systemic state, can exponentially increase the risk of acute CV events that are likely to be precipitated by acute variations in air pollution exposure. Notably, the investigators recently demonstrated that the exposure to higher concentrations of air pollutants (especially PM2.5) is associated with the presence of vulnerable plaque features and with plaque rupture as a mechanism of coronary instability assessed by optical coherence tomography (OCT) and, moreover, with an enhanced systemic and plaque inflammatory activation. In addition, the investigators also demonstrated that a higher exposure to PM2.5 and PM10 in patients with myocardial ischemia and non-obstructive coronary artery disease is associated with coronary vasomotor abnormalities, and PM2.5 is an independent risk factor for the occurrence of epicardial spasm and MINOCA as clinical presentation.

Of interest, even though the pathogenetic mechanism of air pollution are likely to predispose to the occurrence as well as to mediate a worse clinical presentation and outcome of TTS, the relationship between air pollution and the risk of TTS as well as its clinical course has never been assessed. Furthermore, given the poor understanding of the underlying pathophysiology, there is a lack of evidence-based prevention strategies as well as interventions to reduce the incidence as well as the acute complications of TTS.

Upon this background, the investigators hypothesized that:

1. the exposure to higher levels of air pollutants in the days (short-term exposure) or years (long-term exposure) before the TTS onset could be considered as a risk factor for the occurrence of TTS;
2. the exposure to higher levels of air pollutants in the days (short-term exposure) or years (long-term exposure) before the TTS onset could be associated with a worse clinical course in terms of in-hospital complications and mortality;
3. the exposure to higher levels of air pollutants in the days (short-term exposure) or years (long-term exposure) before the TTS onset could be associated with a worse prognosis at follow-up in terms of major adverse cardiovascular events (MACE) and/or TTS recurrence.

In this context, as largely reported throughout the last ten years, time-stratified case-crossover studies represent the best model strategy. In fact, in this study design, instead of comparing exposure between people experiencing a TTS (case) and people who did not (control), pollutant concentrations before TTS diagnosis (case period) were compared with other randomly selected periods, when the subject has not experienced TTS yet (control periods). As such, each patient represents its own control. Hence, time-independent confounders, such as age, comorbidities, and smoking status are controlled by the case-crossover study design, whilst variables that change between case and control time periods are possible confounders (e.g., weather, temperature …). Stratifying by year and month is adequate for most studies and can be done as well by day of the week and temperature.

Primary objective

The primary objective of the study is to assess the relationship between either short-term or long-term exposure to increased levels of air pollutants (PM10, PM2.5, O3, NO2, benzene [C6H6], SO2 e CO) and onset of TTS.

Secondary objectives

* To assess the relationship between either short-term or long-term exposure to increased levels of air pollutants (PM10, PM2.5, O3, NO2, benzene [C6H6], SO2 e CO) and a higher rate of in-hospital complications in patients with TTS.
* To assess the relationship between either a short-term or long-term exposure to increased levels of air pollutants (PM10, PM2.5, O3, NO2, C6H6, SO2 e CO) and a worse clinical outcome at follow-up in patients with TTS.

Study design

Ambispective observational case-crossover pilot study.

Study duration

The study will last 48 months from the approval of the present protocol by the local ethics committee. Enrolment will last 18 months, which will serve also to retrieve the retrospective data from the internal archives. The follow-up period will last 24 months and 6 will be dedicated to the data analysis and interpretation and drafting of scientific reports.

Air pollution data collection

The exposure of patients to air pollution compounds in the two years prior to the occurrence of TTS will be analysed. The investigators will assess: PM10, PM2.5, O3, NO2, C6H6, SO2 e CO. Residential addresses will be obtained from medical records. Annual average 24-h of pollutants levels will be measured matching each individual's home address, obtained through hospital file archive, and the "ArpaLazio" website (http://www.arpalazio.net/main/aria/sci/basedati/chimici/chimici.php). This website provides the concentration values of the following pollutants monitored by the regional automatic network since 1999 and are available for download, expressed as a concentration in micrograms per cubic meter (µg/m3): NO, NO2, NOx, PM10, PM2.5, O3, CO, C6H6, SO2. Hourly data are available for all gaseous pollutants, while the levels of PM10 and PM2.5 are expressed on a daily basis. In addition to the elementary data, the following standard calculations are available: daily averages, typical day, monthly averages and annual averages. The control units are localizable by latitude and longitude coordinates (Sampling Point of Latitude and Longitude) expressed in decimal degrees (DD) and approximated up to the 15th decimal digit, as well as uniquely identifiable by an alphanumeric code (Station Location ID). Data will be obtained from the air quality monitor closest to each participant's residence that was active for the entire year, and short-term (daily and weekly) and long-term (annual) air pollution exposure will be quantified as daily, weekly, and annual average 24-h pollutants level of measurements before TTS. In particular, daily exposure will be assessed as the average 24-h exposure to pollutants the day of TTS onset (0-day lag time between exposure and TTS), the day before (1-day lag time between exposure and TTS), 2 days before (2-day lag time between exposure and TTS), 3 days before (3-day lag time between exposure and TTS), 4 days before (4-day lag time between exposure and TTS), 5 days before (5-day lag time between exposure and TTS), 6 days before (6-day lag time between exposure and TTS) and 7 days before (7-day lag time between exposure and TTS). Similarly, weekly exposure will be assessed as the average 24-h exposure to pollutants the week of TTS onset (0-week lag time between exposure and TTS), the two week before (1-week lag time between exposure and TTS), the three weeks before (2-week lag time between exposure and TTS), and the four week before (3-week lag time between exposure and TTS). Finally, long-term exposure will be assessed as the annual average 24-h pollutants level of measurements of 2 years before TTS. Of note, this methodology to assess air pollution has been extensively validated and used in previous studies. Only patients with 2 years or more of available data on air pollution exposure prior to TTS will be included.

Sample size calculation

To the best of our knowledge, there is no previous literature focusing on air pollutants effects in Takotsubo syndrome (TTS), hence this reflects as a pilot study. As such, no formal sample size calculation is needed. Common rules of thumb for pilot studies by Browne (1995) refer to 30 subjects as a minimum sample size. Based on data retrievable from the archives since 2016 and on an estimated 30 subjects/year diagnosed with TTS at our Unit, the investigators plan to enroll 250 patients in 18 months, which is consistent with the sample size simulation study for case cross-over studies with Dupont's formula, which would imply a sample of at least 195 subjects.

Statistical analysis

The sample will be described in its demographic, anthropometric, clinical, and instrumental, variables through descriptive statistical techniques. In-hospital mortality will be defined as the number of actual (observed) deaths over the total of patients enrolled. In depth, qualitative variables will be expressed by absolute and relative percentage frequencies. Quantitative variables, indeed, will be reported either as mean and standard deviation (SD) or median and interquartile range (IQR), respectively in the case they were normally or not normally distributed. Their distribution will be previously assessed by the Shapiro-Wilk test.

Multiple imputation will be applied to handle missing data, by "imputeR" R package, by using Lasso regression methods centered on the mean for what concerns quantitative variables, whilst classification trees strategy centered on the mode, i.e. the most frequent class, will be applied don qualitative data.

Between groups differences in the demographic, clinical and laboratory features will be assessed by the Chi Square or the Fisher's exact test as for qualitative variables (with Freeman-Halton's extension when appropriate). Differences in the quantitative variables will be instead evaluated either by the Student's t test or the Mann- Withney U test, according to their distribution. Between-groups most significant differences will be further graphically represented by means of "violin plots" drawn with the aid of the R packages "ggstatsplot", "ggpubr" and "ggplot2".

This study will use a time-stratified design to control for time trend and other short-term varying confounders like weather and temperature, as it compares exposure levels between same weekdays/ within each month of each year. Exposure on days where TTS occurred (case days) will be compared with the exposure on days where TTS did not occur (control days). Control days will be chosen on the same day of the week earlier and later in the same month in the same year. Daily TTS counts approximately follow Poisson distribution, hence a linear model of conditional Poisson regression with time-stratified case-crossover design will be fitted to estimate the short- and long-term exposure of air pollutants and TTS risk, applying as potential confounders' parameters such as temperature and weather. Relative Risk (RR) and 95% confidence intervals (CIs) will be estimated based on the per 1 μg/m3 increase of air levels. In the exploratory analysis, the natural cubic splines with three degrees of freedom for temperature, relative humidity and weather will be introduced in new models to examine the nonlinear effect (i.e. the potential confounding by meteorological conditions) and Akaike's Information Criterion will be used to choose the best model. Relative risk increase (RRI) was estimated by RR-1. The RRI in for TTS per 10 μg/m3 increase of PM levels will be calculated as follows: RRI% = exp (β * 10) - 1 * 100%, where β is the exposure-response coefficient from conditional Poisson regression combined under the time-stratified case-crossover design, which refers to a unit increase in PM pollutants. Single-pollutant models will be further implemented to discern the effects of air pollution. When estimating the effects of some potential effect modifiers, time-stratified analyses will be further provided, linking with various subgroups (e.g., by season (warm season: April-September, and cold season: October-March), applying the above analyses for these subgroups. The statistic differences from stratified analyses (e.g., the difference between male and female) will be estimated by Z-test. The same model will be applied also on secondary endpoints of hospitalization rates and MACEs. All analysis will be conducted using R version 4.0.4 with gnm package for conditional Poisson regression combined under the time-stratified case-crossover design.

All statistical tests with p values of < 0.05 will be considered as statistically significant. P-values between 0.05 and 0.10 will be also reported as suggestive. All analyses will be performed by using R software (v. 4.2.0, R Core Team, Vienna, Austria, 2022).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of TTS.
* Available data for short-term and/or long-term exposure to air pollutants (see below).
* Written informed consent to participate.

Exclusion Criteria:

* Age <18 years.
* Not available data for short-term and/or long-term exposure to air pollutants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll all patients admitted to the Department of Cardiovascular Sciences of Fondazione Policlinico Universitario A. Gemelli IRCCS with a diagnosis of TTS. TTS will be diagnosed based on the most recent InterTAK Diagnostic Criteria (31). Myocarditis will be excluded based on clinical presentation (e.g.: previous flu-like symptoms, increased inflammatory biomarkers) and confirmed by cardiac magnetic resonance. All prospectively enrolled patients will provide written informed consent to participate. We will further include all patients with a confirmed TTS diagnosis made between January 2016 and end of October 2022 (hypothetical beginning of prospective phase).
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Association between levels of PM10 air pollutant and TTS | Up to 30 days
  To assess whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant PM10, expressed as a concentration in micrograms per cubic meter (µg/m3) could be associated with TTS.
Association between levels of PM2.5 air pollutant and TTS | Up to 30 days
  To assess whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant PM2.5, expressed as a concentration in micrograms per cubic meter (µg/m3) could be associated with TTS.
Association between levels of O3 air pollutant and TTS | Up to 30 days
  To evaluate whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutants O3, expressed as concentration in micrograms per cubic meter (µg/m3), could be associated with TTS.
Association between levels of NO2 air pollutant and TTS | Up to 30 days
  To assess whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutants NO2, expressed as a concentration in micrograms per cubic meter (µg/m3) could be associated with TTS.
Association between levels of benzene [C6H6] air pollutant and TTS | Up to 30 days
  To assess whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant benzene [C6H6], expressed as a concentration in micrograms per cubic meter (µg/m3) could be associated with TTS.
Association between levels of SO2 air pollutant and TTS | Up to 30 days
  To assess whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutants SO2, expressed as a concentration in micrograms per cubic meter (µg/m3) could be associated with TTS.
Association between levels of CO air pollutant and TTS | Up to 30 days
  To assess whether short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutants CO, expressed as a concentration in micrograms per cubic meter (µg/m3) could be associated with TTS.

SECONDARY OUTCOMES:
Association between levels of PM10 air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant PM10 could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of PM2.5 air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant PM2.5 could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of O3 air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant O3 could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of NO2 air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant NO2 could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of benzene [C6H6] air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant benzene [C6H6] could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of SO2 air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant SO2 could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of CO air pollutant and in-hospital complications | Up to 30 days
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of air pollutant CO could be associated with a higher rate of in-hospital complications (defined as the necessity of inotropic drugs, necessity of temporary ventricular support, necessity of mechanical ventilation, ventricular arrhythmias, new-onset FA, stroke/TIA, in-hospital death) in patients with TTS.
Association between levels of PM10 air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of PM10 air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.
Association between levels of PM2.5 air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of PM2.5 air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.
Association between levels of O3 air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of O3 air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.
Association between levels of NO2 air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of NO2 air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.
Association between levels of benzene [C6H6] air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of benzene [C6H6] air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.
Association between levels of SO2 air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of SO2 air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.
Association between levels of CO air pollutant and MACE at follow-up | Up to 5 years
  To assess whether a short-term (daily and weekly) or long-term (annual) exposure to increased levels of CO air pollutant could be associated with an increased rate of Major Adverse Cardiovascular Events (MACE) at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rocco A Montone, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghadri JR, Wittstein IS, Prasad A, Sharkey S, Dote K, Akashi YJ, Cammann VL, Crea F, Galiuto L, Desmet W, Yoshida T, Manfredini R, Eitel I, Kosuge M, Nef HM, Deshmukh A, Lerman A, Bossone E, Citro R, Ueyama T, Corrado D, Kurisu S, Ruschitzka F, Winchester D, Lyon AR, Omerovic E, Bax JJ, Meimoun P, Tarantini G, Rihal C, Y-Hassan S, Migliore F, Horowitz JD, Shimokawa H, Luscher TF, Templin C. International Expert Consensus Document on Takotsubo Syndrome (Part I): Clinical Characteristics, Diagnostic Criteria, and Pathophysiology. Eur Heart J. 2018 Jun 7;39(22):2032-2046. doi: 10.1093/eurheartj/ehy076. PMID 29850871
- [Background] Lyon AR, Citro R, Schneider B, Morel O, Ghadri JR, Templin C, Omerovic E. Pathophysiology of Takotsubo Syndrome: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Feb 23;77(7):902-921. doi: 10.1016/j.jacc.2020.10.060. PMID 33602474
- [Background] Santoro F, Nunez Gil IJ, Stiermaier T, El-Battrawy I, Guerra F, Novo G, Guastafierro F, Tarantino N, Novo S, Mariano E, Romeo F, Romeo F, Capucci A, Bahlmann E, Zingaro M, Cannone M, Caldarola P, Marchetti MF, Montisci R, Meloni L, Thiele H, Di Biase M, Almendro-Delia M, Sionis A, Akin I, Eitel I, Brunetti ND. Assessment of the German and Italian Stress Cardiomyopathy Score for Risk Stratification for In-hospital Complications in Patients With Takotsubo Syndrome. JAMA Cardiol. 2019 Sep 1;4(9):892-899. doi: 10.1001/jamacardio.2019.2597. PMID 31389988
- [Background] Gili S, Cammann VL, Schlossbauer SA, Kato K, D'Ascenzo F, Di Vece D, Jurisic S, Micek J, Obeid S, Bacchi B, Szawan KA, Famos F, Sarcon A, Levinson R, Ding KJ, Seifert B, Lenoir O, Bossone E, Citro R, Franke J, Napp LC, Jaguszewski M, Noutsias M, Munzel T, Knorr M, Heiner S, Katus HA, Burgdorf C, Schunkert H, Thiele H, Bauersachs J, Tschope C, Pieske BM, Rajan L, Michels G, Pfister R, Cuneo A, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Banning A, Cuculi F, Kobza R, Fischer TA, Vasankari T, Airaksinen KEJ, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Empen K, Felix SB, Delmas C, Lairez O, El-Battrawy I, Akin I, Borggrefe M, Gilyarova E, Shilova A, Gilyarov M, Horowitz JD, Kozel M, Tousek P, Widimsky P, Winchester DE, Ukena C, Gaita F, Di Mario C, Wischnewsky MB, Bax JJ, Prasad A, Bohm M, Ruschitzka F, Luscher TF, Ghadri JR, Templin C. Cardiac arrest in takotsubo syndrome: results from the InterTAK Registry. Eur Heart J. 2019 Jul 1;40(26):2142-2151. doi: 10.1093/eurheartj/ehz170. PMID 31098611
- [Background] Lyon AR, Bossone E, Schneider B, Sechtem U, Citro R, Underwood SR, Sheppard MN, Figtree GA, Parodi G, Akashi YJ, Ruschitzka F, Filippatos G, Mebazaa A, Omerovic E. Current state of knowledge on Takotsubo syndrome: a Position Statement from the Taskforce on Takotsubo Syndrome of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2016 Jan;18(1):8-27. doi: 10.1002/ejhf.424. Epub 2015 Nov 9. PMID 26548803
- [Background] Ortak J, Khattab K, Barantke M, Wiegand UK, Bansch D, Ince H, Nienaber CA, Bonnemeier H. Evolution of cardiac autonomic nervous activity indices in patients presenting with transient left ventricular apical ballooning. Pacing Clin Electrophysiol. 2009 Mar;32 Suppl 1:S21-5. doi: 10.1111/j.1540-8159.2008.02221.x. PMID 19250097
- [Background] Suzuki H, Matsumoto Y, Kaneta T, Sugimura K, Takahashi J, Fukumoto Y, Takahashi S, Shimokawa H. Evidence for brain activation in patients with takotsubo cardiomyopathy. Circ J. 2014;78(1):256-8. doi: 10.1253/circj.cj-13-1276. Epub 2013 Nov 28. PMID 24284957
- [Background] Hiestand T, Hanggi J, Klein C, Topka MS, Jaguszewski M, Ghadri JR, Luscher TF, Jancke L, Templin C. Takotsubo Syndrome Associated With Structural Brain Alterations of the Limbic System. J Am Coll Cardiol. 2018 Feb 20;71(7):809-811. doi: 10.1016/j.jacc.2017.12.022. No abstract available. PMID 29447745
- [Background] Galiuto L, De Caterina AR, Porfidia A, Paraggio L, Barchetta S, Locorotondo G, Rebuzzi AG, Crea F. Reversible coronary microvascular dysfunction: a common pathogenetic mechanism in Apical Ballooning or Tako-Tsubo Syndrome. Eur Heart J. 2010 Jun;31(11):1319-27. doi: 10.1093/eurheartj/ehq039. Epub 2010 Mar 9. PMID 20215125
- [Background] De Caterina AR, Leone AM, Galiuto L, Basile E, Fedele E, Paraggio L, De Maria GL, Porto I, Niccoli G, Burzotta F, Trani C, Rebuzzi AG, Crea F. Angiographic assessment of myocardial perfusion in Tako-Tsubo syndrome. Int J Cardiol. 2013 Oct 12;168(5):4717-22. doi: 10.1016/j.ijcard.2013.07.172. Epub 2013 Jul 25. PMID 23948116
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] Landrigan PJ, Fuller R, Acosta NJR, Adeyi O, Arnold R, Basu NN, Balde AB, Bertollini R, Bose-O'Reilly S, Boufford JI, Breysse PN, Chiles T, Mahidol C, Coll-Seck AM, Cropper ML, Fobil J, Fuster V, Greenstone M, Haines A, Hanrahan D, Hunter D, Khare M, Krupnick A, Lanphear B, Lohani B, Martin K, Mathiasen KV, McTeer MA, Murray CJL, Ndahimananjara JD, Perera F, Potocnik J, Preker AS, Ramesh J, Rockstrom J, Salinas C, Samson LD, Sandilya K, Sly PD, Smith KR, Steiner A, Stewart RB, Suk WA, van Schayck OCP, Yadama GN, Yumkella K, Zhong M. The Lancet Commission on pollution and health. Lancet. 2018 Feb 3;391(10119):462-512. doi: 10.1016/S0140-6736(17)32345-0. Epub 2017 Oct 19. No abstract available. PMID 29056410
- [Background] Brauer M, Casadei B, Harrington RA, Kovacs R, Sliwa K; WHF Air Pollution Expert Group. Taking a Stand Against Air Pollution-The Impact on Cardiovascular Disease: A Joint Opinion from the World Heart Federation, American College of Cardiology, American Heart Association, and the European Society of Cardiology. J Am Coll Cardiol. 2021 Apr 6;77(13):1684-1688. doi: 10.1016/j.jacc.2020.12.003. Epub 2021 Jan 28. PMID 33518378
- [Background] Lelieveld J, Klingmuller K, Pozzer A, Poschl U, Fnais M, Daiber A, Munzel T. Cardiovascular disease burden from ambient air pollution in Europe reassessed using novel hazard ratio functions. Eur Heart J. 2019 May 21;40(20):1590-1596. doi: 10.1093/eurheartj/ehz135. PMID 30860255
- [Background] Franck U, Odeh S, Wiedensohler A, Wehner B, Herbarth O. The effect of particle size on cardiovascular disorders--the smaller the worse. Sci Total Environ. 2011 Sep 15;409(20):4217-21. doi: 10.1016/j.scitotenv.2011.05.049. Epub 2011 Aug 10. PMID 21835436
- [Background] Turner MC, Jerrett M, Pope CA 3rd, Krewski D, Gapstur SM, Diver WR, Beckerman BS, Marshall JD, Su J, Crouse DL, Burnett RT. Long-Term Ozone Exposure and Mortality in a Large Prospective Study. Am J Respir Crit Care Med. 2016 May 15;193(10):1134-42. doi: 10.1164/rccm.201508-1633OC. PMID 26680605
- [Background] Rajagopalan S, Landrigan PJ. Pollution and the Heart. N Engl J Med. 2021 Nov 11;385(20):1881-1892. doi: 10.1056/NEJMra2030281. No abstract available. PMID 34758254
- [Background] Rajagopalan S, Al-Kindi SG, Brook RD. Air Pollution and Cardiovascular Disease: JACC State-of-the-Art Review. J Am Coll Cardiol. 2018 Oct 23;72(17):2054-2070. doi: 10.1016/j.jacc.2018.07.099. PMID 30336830
- [Background] Bevan GH, Al-Kindi SG, Brook RD, Munzel T, Rajagopalan S. Ambient Air Pollution and Atherosclerosis: Insights Into Dose, Time, and Mechanisms. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):628-637. doi: 10.1161/ATVBAHA.120.315219. Epub 2020 Dec 17. PMID 33327745
- [Background] Al-Kindi SG, Brook RD, Biswal S, Rajagopalan S. Environmental determinants of cardiovascular disease: lessons learned from air pollution. Nat Rev Cardiol. 2020 Oct;17(10):656-672. doi: 10.1038/s41569-020-0371-2. Epub 2020 May 7. PMID 32382149
- [Background] Brook RD, Rajagopalan S, Pope CA 3rd, Brook JR, Bhatnagar A, Diez-Roux AV, Holguin F, Hong Y, Luepker RV, Mittleman MA, Peters A, Siscovick D, Smith SC Jr, Whitsel L, Kaufman JD; American Heart Association Council on Epidemiology and Prevention, Council on the Kidney in Cardiovascular Disease, and Council on Nutrition, Physical Activity and Metabolism. Particulate matter air pollution and cardiovascular disease: An update to the scientific statement from the American Heart Association. Circulation. 2010 Jun 1;121(21):2331-78. doi: 10.1161/CIR.0b013e3181dbece1. Epub 2010 May 10. PMID 20458016
- [Background] Yang S, Lee SP, Park JB, Lee H, Kang SH, Lee SE, Kim JB, Choi SY, Kim YJ, Chang HJ. PM2.5 concentration in the ambient air is a risk factor for the development of high-risk coronary plaques. Eur Heart J Cardiovasc Imaging. 2019 Dec 1;20(12):1355-1364. doi: 10.1093/ehjci/jez209. PMID 31410457
- [Background] Araujo JA, Barajas B, Kleinman M, Wang X, Bennett BJ, Gong KW, Navab M, Harkema J, Sioutas C, Lusis AJ, Nel AE. Ambient particulate pollutants in the ultrafine range promote early atherosclerosis and systemic oxidative stress. Circ Res. 2008 Mar 14;102(5):589-96. doi: 10.1161/CIRCRESAHA.107.164970. Epub 2008 Jan 17. PMID 18202315
- [Background] Montone RA, Camilli M, Russo M, Termite C, La Vecchia G, Iannaccone G, Rinaldi R, Gurgoglione F, Del Buono MG, Sanna T, Trani C, Liuzzo G, Crea F, Niccoli G. Air Pollution and Coronary Plaque Vulnerability and Instability: An Optical Coherence Tomography Study. JACC Cardiovasc Imaging. 2022 Feb;15(2):325-342. doi: 10.1016/j.jcmg.2021.09.008. Epub 2021 Oct 13. PMID 34656488
- [Background] Camilli M, Russo M, Rinaldi R, Caffe A, La Vecchia G, Bonanni A, Iannaccone G, Basile M, Vergallo R, Aurigemma C, Trani C, Niccoli G, Crea F, Montone RA. Air Pollution and Coronary Vasomotor Disorders in Patients With Myocardial Ischemia and Unobstructed Coronary Arteries. J Am Coll Cardiol. 2022 Nov 8;80(19):1818-1828. doi: 10.1016/j.jacc.2022.08.744. Epub 2022 Aug 29. PMID 36049556
- [Background] Collart P, Coppieters Y, Mercier G, Massamba Kubuta V, Leveque A. Comparison of four case-crossover study designs to analyze the association between air pollution exposure and acute myocardial infarction. Int J Environ Health Res. 2015;25(6):601-13. doi: 10.1080/09603123.2014.1003037. Epub 2015 Feb 4. PMID 25650956
- [Background] Rich DQ, Kipen HM, Zhang J, Kamat L, Wilson AC, Kostis JB. Triggering of transmural infarctions, but not nontransmural infarctions, by ambient fine particles. Environ Health Perspect. 2010 Sep;118(9):1229-34. doi: 10.1289/ehp.0901624. Epub 2010 Apr 30. PMID 20435544
- [Background] Gardner B, Ling F, Hopke PK, Frampton MW, Utell MJ, Zareba W, Cameron SJ, Chalupa D, Kane C, Kulandhaisamy S, Topf MC, Rich DQ. Ambient fine particulate air pollution triggers ST-elevation myocardial infarction, but not non-ST elevation myocardial infarction: a case-crossover study. Part Fibre Toxicol. 2014 Jan 2;11:1. doi: 10.1186/1743-8977-11-1. PMID 24382024
- [Background] Janes H, Sheppard L, Lumley T. Case-crossover analyses of air pollution exposure data: referent selection strategies and their implications for bias. Epidemiology. 2005 Nov;16(6):717-26. doi: 10.1097/01.ede.0000181315.18836.9d. PMID 16222160
- [Background] Jaakkola JJ. Case-crossover design in air pollution epidemiology. Eur Respir J Suppl. 2003 May;40:81s-85s. doi: 10.1183/09031936.03.00402703. PMID 12762580
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Dharmarajan S, Lee JY, Izem R. Sample size estimation for case-crossover studies. Stat Med. 2019 Mar 15;38(6):956-968. doi: 10.1002/sim.8030. Epub 2018 Nov 5. PMID 30397907